CLINICAL TRIAL: NCT05400902
Title: Hepatic Arterial Infusion Chemotherapy Combined With Sintilimab and Bevacizumab in the Treatment of Unresectable Intrahepatic Cholangiocarcinoma: A Prospective, Single-Center, Phase II Study
Brief Title: HAIC Combined With Sintilimab and Bevacizumab for Unresectable Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Binkui Li (Other)
Responsible Party: Sponsor-Investigator, Binkui Li, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-233-01
Record Dates: First submitted 2022-05-28; First posted 2022-06-02 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Hepatic Arterial Infusion Chemotherapy; Sintilimab; Bevacizumab
MeSH Terms: conditions — Cholangiocarcinoma | interventions — tislelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC Combined with Sintilimab and Bevacizumab (Experimental)
  Interventions: Drug: HAIC Combined with Tislelizumab and Apatinib

INTERVENTIONS:
Drug: HAIC Combined with Tislelizumab and Apatinib — Hepatic Arterial Infusion Chemotherapy: FOLFOX6 regimen was infused with chemotherapy drugs: oxaliplatin 130 mg/m2 infusion for 2 hours, folinate calcium 400 mg/m2 infusion for 2 hours, 5-fluorouracil 400 mg/m2 arterial infusion for 10 minutes, 5-fluorouracil 1200 mg/m2 infusion for 23 hours. Every 3 weeks, no more than 4 cycles of HAIC treatment.
  Sintilimab and Bevacizumab treatment: start at 0-3 days after the end of hepatic arterial infusion chemotherapy: Sintilimab 200 mg ivdrip, Q3W; Bevacizumab 15 mg/kg ivdrip, Q3W

SUMMARY:
Primary liver cancer is the sixth most common cancer worldwide, including hepatocellular carcinoma and intrahepatic cholangiocarcinoma, of which intrahepatic cholangiocarcinoma accounts for 10%-15%. Surgical resection is the only curative method for ICC, but most patients are diagnosed at an advanced stage, and only 15% of patients can undergo surgical resection. In locally advanced ICC patients without distant metastases, although the tumor was initially assessed as unresectable, these patients may have the opportunity for surgical resection after reducing the size tumor lesion and increasing the remnant liver volume through conversion therapy. The current standard first-line treatment for unresectable ICC is gemcitabine combined with cisplatin, with a median overall survival of only 11.7 months and an ORR of 26.1%. In view of the poor effect of the standard chemotherapy regimen, the NCCN guidelines recommend that patients could participate in clinical study. Hepatic arterial infusion chemotherapy can increase the local blood drug concentration and improve the tumor regression rate. By reducing the dose of systemic chemotherapy drugs concentration, the incidence of adverse reactions can be reduced. Hepatic arterial infusion chemotherapy may be a better choice for locally advanced intrahepatic cholangiocarcinoma. PD-1 immunotherapy combined with targeted therapy is expected to improve the prognosis of patients with intrahepatic cholangiocarcinoma. This study investigates the safety and efficacy of hepatic arterial infusion chemotherapy combined with sintilimab and bevacizumabin the treatment of unresectable ICC.

ELIGIBILITY:
Inclusion Criteria:

* ICC diagnosed by imaging examination (CT or MRI) and pathology;
* ICC patient without any previous tumor treatment
* The tumor was assessed as unresectable by two liver surgeons. Any of the following conditions: (1) Residual liver volume less than 30-40%; (2) Not possible for R0 radical resection; (3) Tumor invades the portal vein, hepatic artery and bile duct, and the normal residual liver cannot be guaranteed blood supply and bile drainage; the tumor involves the hepatic veins and cannot preserve at least one vein.
* At least one assessable intrahepatic lesion;
* ECOG PS score 0-1;
* Child-Pugh class A;
* Life expectancy is at least 3 months;
* Age between 18 and 75 years old;
* Baseline laboratory tests meet the following criteria:

Neutrophils ≥1.5×10^9/L White blood cells ≥3.0×10^9/L Platelets ≥75×10^9/L Hemoglobin ≥80g/L Serum ALT, AST ≤ 3 x upper limit of normal (ULN) Serum creatinine ≤ 1.5 x ULN INR < 1.5, or prothrombin time < ULN+4 seconds Albumin ≥30g/L Total bilirubin ≤ 3 x upper limit of normal (ULN)

Exclusion Criteria:

* Distant metastasis;
* Refused to receive PD-1 inhibitor and apatinib treatment;
* Any of the following conditions within the first 12 months of the study: myocardial infarction, severe/unstable angina, coronary artery bypass grafting, congestive heart failure, cerebrovascular accident (including transient ischemic attack), Pulmonary embolism; ongoing: arrhythmia grade ≥2 according to NCI-CTCAE criteria, QTc prolongation (>450 ms in men, >470 ms in women);
* Renal insufficiency requires peritoneal dialysis or hemodialysis;
* Serious dysfunction of other important organs;
* A second primary malignant tumor was diagnosed in the past;
* Known or new evidence of brain or leptomeningeal lesions;
* Hemophilia or bleeding tendency, who are taking anticoagulation therapy such as coumarin derivatives in therapeutic doses;
* Pregnant or lactating women, all female patients of childbearing potential must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative;
* History of previous organ transplantation;
* Known HIV infection;
* Allergy to chemotherapy drugs;
* Patients with other serious acute or chronic physical or psychiatric diseases or abnormal laboratory tests that may increase the risk associated with participating in the study, or may interfere with the interpretation of the study results or the investigators consider unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 12 months
  The objective response rate was calculated according to the RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  defined as the time from the start of enrollment to the time of tumor progression (PD) or death or last follow-up on imaging.
Disease Control Rate | 12 months
  According to the RECIST 1.1 standard, complete remission + partial remission + disease control rate were calculated.
Conversion rate to resection | 12 months
  Defined as the rate of surgical resection among all enrolled patients.
Overall Survival time | 12 months
  Defined as the time from enrollment until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No